CLINICAL TRIAL: NCT03264885
Title: Randomized Controlled Trial Evaluating an Incentive-based Community Eye-care Programme for Elderly With Visual Impairment
Brief Title: Randomized Controlled Trial Evaluating an Incentive-based Community Eye-care Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R1102/4/2014
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2017-08

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The usual stand of care (UC) after community eye screening was to provide a GP referral letter and advice to attend a tertiary eye care facility most accessible to them
- Incentive Care (Other): In addition to the UC, those assigned to the ICS also received social and financial support to incentivise and improve compliance. All ICS participants were assisted with scheduling their tertiary care appointments, given telephone reminders, provided once-off transportation allowance and subsidy for their first tertiary eye-care consultation - while participants with mobility issues were assisted by volunteers.
  Interventions: Other: Incentive Care

INTERVENTIONS:
Other: Incentive Care — ICS is a novel intervention that incorporates patient education, social support, and financial assistance to assist individuals.
  Arms: Incentive Care

SUMMARY:
Elderly with visual impairment (VI) who undergo community eye screening often do not attend tertiary follow-up even if significant eye diseases are detected. Investigators evaluate an incentive-care scheme (ICS) to improve the attendance rates of tertiary eye-care visits of participants following community eye screening.

DETAILED DESCRIPTION:
A randomized controlled study individuals with VI with baseline visual acuity (VA) and vision-related quality of life (VRQoL) assessed in the community. Participants were randomised to either receiving ICS or usual care (UC). ICS is a novel intervention that incorporates patient education, social support, and financial assistance to assist individuals. Participants in UC received a standard GP referral letter advising them to seek further care. Our main outcome measure was compliance to tertiary eye-care referral. Our secondary outcome measure was VA and VRQoL assessed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* the ability to speak English and/or Mandarin, have adequate hearing with/without hearing aids to respond to normal conversation, not currently undergoing regular assessment/care with an ophthalmologist (at least yearly), have the ability to undergo visual acuity testing and provide reliable results, and visual acuity of 6/12 or worse in either eye after best correction

Exclusion Criteria:

* refused informed consent and any other contraindication(s) as indicated by the general practitioner responsible for the participant

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Compliance to Tertiary Care Follow-up | 3 months
  Percentage of participants who attended follow-up

SECONDARY OUTCOMES:
Visual Acuity | 3 months
  Vision checked on Snellen chart

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Ang, Principal Investigator — SNEC

IPD SHARING:
Plan to Share IPD: No
Data will not be available to other researchers